CLINICAL TRIAL: NCT02563834
Title: A Novel Positron Emission Tomography (PET) Approach to Measuring Myocardial Metabolism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 10100002643; R21DK071142 (NIH)
Record Dates: First submitted 2015-09-29; First posted 2015-09-30 (Estimated); Results first posted 2016-08-31 (Estimated); Last update posted 2016-08-31 (Estimated); Status verified 2016-08

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Sodium Chloride; Insulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Saline (Experimental): Studies will be performed on one day under fasting conditions, using a saline infusion. All subjects will receive infusions of radiolabeled acetate and radiolabeled thiapalmitate tracer (16-18-F-fluoro-4-thiapalmitate).
  Interventions: Drug: thiapalmitate tracer; Drug: Saline
- Insulin Clamp (Experimental): Studies will be performed on a separate day under fasting conditions, using an insulin infusion to achieve steady state insulin/glucose clamp conditions. Studies will be performed on one day under fasting conditions, using a saline infusion. All subjects will receive infusions of radiolabeled acetate and radiolabeled thiapalmitate tracer (16-18-F-fluoro-4-thiapalmitate).
  Interventions: Drug: thiapalmitate tracer; Drug: Insulin

INTERVENTIONS:
Drug: thiapalmitate tracer — Radiolabeled tracer infusion; occurs in all treatment arms
  Other Names: 16- 18-F-fluoro-4-thiapalmitate
Drug: Saline — Saline infusion for control
  Arms: Saline
Drug: Insulin — Insulin infusion for insulin/glucose clamp procedure
  Arms: Insulin Clamp

SUMMARY:
Studies of myocardial fuel selection using a novel palmitate-based PET probe

DETAILED DESCRIPTION:
A novel Positron Emission Tomography (PET) probe, 16- 18-F-fluoro-4-thiapalmitate, will be used to evaluate myocardial atty acid uptake. Studies will be done in humans with type 2 diabetes mellitus, and in controls. Studies will take place on 2 separate days, under fasting conditions and under insulin clamp conditions.

ELIGIBILITY:
Inclusion Criteria:

* Lean:

  * BMI<25 kg/m2
  * normal glucose tolerance by 75g oral glucose tolerance test
* Type 2 diabetes mellitus:

  * BMI >25 kg/m2
  * previously diagnosed type 2 diabetes mellitus
  * on oral and/or injected insulin treatment.

Exclusion Criteria:

* Lean:

  *Use of any chronic medications
* Type 2 diabetes mellitus

  * known microvascular disease
  * known coronary or other macro vascular disease
  * use of PPARgamma class antidiabetic agents within 6 months

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2007-01; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kieren J Mather, MD, Principal Investigator — Indiana University
Locations (1):
- Indiana University Hospital GCRC, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Mather KJ, Hutchins GD, Perry K, Territo W, Chisholm R, Acton A, Glick-Wilson B, Considine RV, Moberly S, DeGrado TR. Assessment of myocardial metabolic flexibility and work efficiency in human type 2 diabetes using 16-[18F]fluoro-4-thiapalmitate, a novel PET fatty acid tracer. Am J Physiol Endocrinol Metab. 2016 Mar 15;310(6):E452-60. doi: 10.1152/ajpendo.00437.2015. Epub 2016 Jan 5. PMID 26732686

RESULTS

PARTICIPANT FLOW:
Groups:
- Lean Control: Studies will be performed on 2 separate days under fasting conditions, using a saline infusion on Day 1 and insulin infusion on Day 2. All subjects will receive infusions of radiolabeled acetate and radiolabeled thiapalmitate tracer (16-18-F-fluoro-4-thiapalmitate) on both study days.
  thiapalmitate tracer: Radiolabeled tracer infusion; occurs in all treatment arms
  Saline: Saline infusion for control
- Type 2 DM: Studies will be performed on 2 separate days under fasting conditions, using a saline infusion on Day 1 and insulin infusion on Day 2. All subjects will receive infusions of radiolabeled acetate and radiolabeled thiapalmitate tracer (16-18-F-fluoro-4-thiapalmitate) on both study days.
  thiapalmitate tracer: Radiolabeled tracer infusion; occurs in all treatment arms
Period: Control (Saline) Infusion (*Day 1)
Arm/Group | Lean Control | Type 2 DM
Started | 10 | 8
Completed | 10 | 8
Not Completed | 0 | 0
Period: Insulin Infusion (*Day 2)
Arm/Group | Lean Control | Type 2 DM
Started | 10 | 8
Completed | 10 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Lean Controls: Lean non-diabetic control participants, taking no regular medications.
- Type 2 Diabetes: Participants with Type 2 diabetes treated with any combination of oral agents and insulin except PPARgamma agonists.
- Total: Total of all reporting groups
Arm/Group | Lean Controls | Type 2 Diabetes | Total
Number analyzed (Participants) | 10 | 8 | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 8 | 18
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.1 (9.0) | 40.4 (9.2) | 36.9 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 5 | 15
  Male | 0 | 3 | 3

OUTCOME MEASURES:

1. Primary Outcome: Myocardial Fatty Acid Uptake Rate
Description: PET measure of fatty acid uptake rate
Time Frame: 4 Hours
Measure: Mean (Standard Error); unit: umol/min/100g
Groups:
- Lean Control - Saline: Studies will be performed on a separate day under fasting conditions, using a saline infusion. All subjects will receive infusions of radiolabeled acetate and radiolabeled thiapalmitate tracer (16-18-F-fluoro-4-thiapalmitate).
  thiapalmitate tracer: Radiolabeled tracer infusion; occurs in all treatment arms
  Saline: Saline infusion for control
- Lean Control - Insulin Clamp: Studies will be performed on a separate day under fasting conditions, using an insulin infusion to achieve steady state insulin/glucose clamp conditions. All subjects will receive infusions of radiolabeled acetate and radiolabeled thiapalmitate tracer (16-18-F-fluoro-4-thiapalmitate).
  thiapalmitate tracer: Radiolabeled tracer infusion; occurs in all treatment arms
  Insulin: Insulin infusion for insulin/glucose clamp procedure
- Type 2 DM - Saline: Studies will be performed on a separate day under fasting conditions, using a saline infusion. All subjects will receive infusions of radiolabeled acetate and radiolabeled thiapalmitate tracer (16-18-F-fluoro-4-thiapalmitate).
  thiapalmitate tracer: Radiolabeled tracer infusion; occurs in all treatment arms
- Type 2 DM - Insulin Clamp: Studies will be performed on a separate day under fasting conditions, using an insulin infusion to achieve steady state insulin/glucose clamp conditions. All subjects will receive infusions of radiolabeled acetate and radiolabeled thiapalmitate tracer (16-18-F-fluoro-4-thiapalmitate).
  thiapalmitate tracer: Radiolabeled tracer infusion; occurs in all treatment arms
Arm/Group | Lean Control - Saline | Lean Control - Insulin Clamp | Type 2 DM - Saline | Type 2 DM - Insulin Clamp
Number analyzed (Participants) | 10 | 10 | 8 | 8
umol/min/100g | 18.492 (3.942) | 2.123 (1.087) | 36.005 (4.408) | 7.8 (1.215)

2. Secondary Outcome: Myocardial Oxidation Rate
Description: PET measure of total oxidation rate
Time Frame: 4 Hours
Measure: Mean (Standard Error); unit: ml/min/100g
Arm/Group | Lean Control - Saline | Lean Control - Insulin Clamp | Type 2 DM - Saline | Type 2 DM - Insulin Clamp
Number analyzed (Participants) | 10 | 10 | 8 | 8
ml/min/100g | 15.006 (0.951) | 19.847 (1.773) | 17.381 (1.064) | 22.940 (2.288)

3. Secondary Outcome: Myocardial Perfusion Rate
Description: PET measure of total myocardial perfusion (blood flow)
Time Frame: 4 Hours
Measure: Mean (Standard Error); unit: ml/min/100g
Arm/Group | Lean Control - Saline | Lean Control - Insulin Clamp | Type 2 DM - Saline | Type 2 DM - Insulin Clamp
Number analyzed (Participants) | 10 | 10 | 8 | 8
ml/min/100g | 39.3 (2.1) | 46.5 (3.3) | 44.2 (2.3) | 49.4 (4.2)

ADVERSE EVENTS:
Arm/Group | Saline | Insulin Clamp
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/18
Other Adverse Events (participants affected / at risk) | 0/18 | 0/18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No